CLINICAL TRIAL: NCT01714349
Title: Restoring Hand Function Using Nerve Transfers in Persons With Spinal Cord Injury
Brief Title: Nerve Transfer After Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTSCI -201208137
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; nerve transfer; tetraplegia; quadriplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Nerve Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nerve Transfer (Experimental): Surgical - Nerve transfers for patients with stable cervical spinal cord injuries
  Interventions: Procedure: Nerve Transfer

INTERVENTIONS:
Procedure: Nerve Transfer — A nerve transfer procedure will be individualized to each patient's functional deficit.

SUMMARY:
Nerve Transfer surgery can provide improved hand function following cervical spinal cord injuries

DETAILED DESCRIPTION:
Current treatment strategies of acute cervical spinal cord injuries remain limited. Treatment options that provide meaningful improvements in patient quality of life and long-term functional independence will provide a significant public health impact.

Specific Aim: Measure the efficacy of nerve transfer surgery in the treatment of patients with complete cervical spinal cord injuries with no hand function. Optimize the efficiency of nerve transfer surgery by evaluating patient outcomes in relation to patient selection and optimal timing the the surgery.

Hypothesis: Peripheral nerve transfers in patients with spinal cord injuries will improve hand function and provide improvement in patient quality of life and functional independence.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Informed Consent Document (ICD) signed by patient
3. Cervical spinal cord injury resulting in arm & hand functional impairment, with at least preserved elbow function
4. International Classification of Surgery of the Hand in Tetraplegia (ICSHT) category 0 - 4
5. Patients with a stable American Spinal Injury Association (ASIA) grade of A, B, or C, or with a diagnosis of central cord syndrome, showing minimal to no evidence of functional improvement in motor examination after at least 6 months of non-operative therapy post-injury
6. Appropriate candidate for nerve transfer study
7. Willing and able to comply with the study protocol
8. < 48 months from injury

Exclusion Criteria:

1. Active infection at the operative site or systemic infection
2. Any return or ongoing clinical recovery of distal motor function within 6 months after injury
3. Physically or mentally compromised
4. Currently undergoing long-term steroid therapy
5. Significant joint contractures and/or limitations in passive range of motion in the arm or hand
6. Active malignancy
7. Systemic disease that would affect the patient's welfare or the research study
8. Pregnant
9. Immunologically suppressed or immunocompromised
10. Significant pain or hypersensitivity
11. Previous or current injury preventing use of tendon transfers to restore upper extremity function
12. Affective disorder of a degree that would make outcome assessment and study participation difficult
13. History of brachial plexus injury or systemic neuropathic process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in upper motor strength | 48 months
  Patients motor strength will be assessed over 48 months of clinical follow-up with conventional manual motor testing

SECONDARY OUTCOMES:
Change in Disabilities of Arm, Shoulder, and Hand (DASH) scores | 48 months
  The change in DASH scores will be followed over time and assessed pre-operatively, 6,12, 18, 24, 36 and 48 months post-operatively.
Change in Short Form 36 (SF-36) scores | 48 months
  The change in SF-36 scores will be followed over time and assessed pre-operatively, 6, 12, 18, 24. 36 and 48 months post-operatively.
Change in Michigan Hand Questionnaire (MHQ) | 48 months
  The change in MHQ will be followed over time and assessed pre-operatively, 6, 12, 18, 24, 36 and 48 months post-operatively.

OTHER OUTCOMES:
Rates of Intraoperative and Post-operative complications | 48 months
  The number of complications within and after the operation.
Effect of timing on surgical intervention | 48 months
  Assess the effect of timing on primary and secondary outcome measures, early (<12 months) vs. (>12 months)
Rate of reoperation | 48 months
  The rate at which a patient needs to be operated on again.
Hand Function, measured by the Sollerman Hand Function Test | 48 months
  The Sollerman Hand Function Test is performed as part of an overall evaluation and assessment by study team Occupational Therapist pre-operatively, post-operatively, and at 6 months, 12 months, 18 months, and 24 months. 36 months and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- See also: Washington University Neurosurgery Home Page — http://www.neurosurgery.wustl.edu